CLINICAL TRIAL: NCT02101775
Title: A Randomized Placebo-Controlled Phase II Trial Comparing Gemcitabine Monotherapy to Gemcitabine in Combination With AZD 1775 (MK 1775) in Women With Recurrent, Platinum Resistant Epithelial Ovarian, Primary Peritoneal, or Fallopian Tube Cancers
Brief Title: Gemcitabine Hydrochloride With or Without WEE1 Inhibitor MK-1775 in Treating Patients With Recurrent Ovarian, Primary Peritoneal, or Fallopian Tube Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NCI-2014-00620; NCI-2014-00620 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PHL-093; NCI 9568; 9568 (Other: University Health Network-Princess Margaret Hospital); 9568 (Other: CTEP); N01CM00032 (NIH); N01CM00038 (NIH); N01CM00071 (NIH); U10CA180821 (NIH); UM1CA186644 (NIH); UM1CA186705 (NIH); NCT02151292 (obsolete NCT alias)
Record Dates: First submitted 2014-03-28; First posted 2014-04-02 (Estimated); Results first posted 2023-09-08 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Ovarian Brenner Tumor; Ovarian Carcinosarcoma; Ovarian Clear Cell Cystadenocarcinoma; Ovarian Endometrioid Adenocarcinoma; Ovarian Mucinous Cystadenocarcinoma; Ovarian Seromucinous Carcinoma; Ovarian Serous Cystadenocarcinoma; Ovarian Serous Surface Papillary Adenocarcinoma; Ovarian Undifferentiated Carcinoma; Recurrent Fallopian Tube Carcinoma; Recurrent Ovarian Carcinoma; Recurrent Primary Peritoneal Carcinoma
MeSH Terms: conditions — Brenner Tumor; Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — adavosertib; Gemcitabine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (WEE1 inhibitor MK-1775, gemcitabine hydrochloride) (Experimental): Patients receive WEE1 inhibitor MK-1775 PO on days 1, 2, 8, 9, 15, and 16 and gemcitabine hydrochloride IV over 30 minutes on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Adavosertib; Drug: Gemcitabine Hydrochloride; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Other: Questionnaire Administration
- Arm II (placebo, gemcitabine hydrochloride) (Active Comparator): Patients receive placebo PO on days 1, 2, 8, 9, 15, and 16 and gemcitabine hydrochloride as patients in Arm I. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Gemcitabine Hydrochloride; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Other: Placebo Administration; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Adavosertib — Given PO
  Other Names: AZD 1775; AZD-1775; AZD1775; MK 1775; MK-1775; MK1775
  Arms: Arm I (WEE1 inhibitor MK-1775, gemcitabine hydrochloride)
Drug: Gemcitabine Hydrochloride — Given IV
  Other Names: dFdCyd; Difluorodeoxycytidine Hydrochloride; Gemcitabine HCI; Gemzar; LY 188011; LY-188011; LY188011
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Other: Placebo Administration — Given PO
  Arms: Arm II (placebo, gemcitabine hydrochloride)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This randomized phase II clinical trial studies how well gemcitabine hydrochloride and WEE1 inhibitor MK-1775 work compared to gemcitabine hydrochloride alone in treating patients with ovarian, primary peritoneal, or fallopian tube cancer that has come back after a period of time. Gemcitabine hydrochloride may prevent tumor cells from multiplying by damaging their deoxyribonucleic acid (DNA, molecules that contain instructions for the proper development and functioning of cells), which in turn stops the tumor from growing. The protein WEE1 may help to repair the damaged tumor cells, so the tumor continues to grow. WEE1 inhibitor MK-1775 may block the WEE1 protein activity and may increase the effectiveness of gemcitabine hydrochloride by preventing the WEE1 protein from repairing damaged tumor cells without causing harm to normal cells. It is not yet known whether gemcitabine hydrochloride with or without WEE1 inhibitor MK-1775 may be an effective treatment for recurrent ovarian, primary peritoneal, or fallopian tube cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the progression free survival (PFS) of subjects with recurrent platinum-resistant ovarian, fallopian tube or primary peritoneal cancer receiving gemcitabine (gemcitabine hydrochloride) in combination with AZD 1775 (MK-1775 [WEE1 inhibitor MK-1775]) compared to subjects receiving gemcitabine in combination with placebo.

SECONDARY OBJECTIVES:

I. To evaluate the objective response by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 of patients receiving gemcitabine combined with AZD 1775 (MK-1775) compared to patients receiving gemcitabine in combination with placebo.

II. To evaluate the Gynecologic Cancer Intergroup (GCIG) cancer antigen (CA)125 response rate of patients receiving gemcitabine combined with AZD 1775 (MK-1775) compared to patients receiving gemcitabine in combination with placebo.

III. To evaluate the overall survival of patients (max 1-year [yr] follow-up) receiving gemcitabine combined with AZD 1775 (MK-1775) compared to patients receiving gemcitabine in combination with placebo.

IV. To evaluate the safety and tolerability of the combination of gemcitabine combined with AZD 1775 (MK-1775) in patients with recurrent, platinum-resistant ovarian, fallopian tube or primary peritoneal cancer.

V. To evaluate tumor protein p53 (TP53) mutations (presence of mutation and type of mutation) as potential predictive factors of benefit (defined as response or progression-free survival [PFS] prolongation) to AZD 1775 (MK-1775) and gemcitabine treatment.

VI. To evaluate p53 protein expression by immunohistochemistry as potential predictive factors of benefit (defined as response or PFS prolongation) to AZD 1775 (MK-1775) and gemcitabine treatment.

TERTIARY OBJECTIVES:

I. To evaluate patient reported outcomes using Patient-Reported Outcomes (PRO)-Common Terminology Criteria for Adverse Events (CTCAE).

II. To evaluate the concordance of TP53 mutations in the tumor specimen and TP53 mutations determined by tagged-amplicon deep sequencing (Tam-Seq) in circulating tumor DNA.

III. To correlate the levels circulating DNA TP53 mutations by Tam-Seq with response.

IV. Validation of phosphorylated-cyclin-dependent cycle 2 (pCDC2) and gamma-H2A histone family, member X (H2AX) in skin and tumor tissue as a pharmacodynamic marker of therapy.

V. To correlate changes in pCDC2 and gamma-H2AX with survival outcomes and response rate.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive WEE1 inhibitor MK-1775 orally (PO) on days 1, 2, 8, 9, 15, and 16 and gemcitabine hydrochloride intravenously (IV) over 30 minutes on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive placebo PO on days 1, 2, 8, 9, 15, and 16 and gemcitabine hydrochloride as patients in Arm I. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6-8 weeks (after the 30-37 day safety visit) for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed epithelial ovarian, primary peritoneal and fallopian tube carcinoma; all histologic subtypes of epithelial ovarian cancer are eligible, but only patients with high grade serous ovarian cancer will be considered for the statistical analysis; non-high grade serous cancers will be allowed in an exploratory cohort
* Patients must be platinum-resistant (platinum-free interval < 6 months) or have platinum-refractory disease as per Gynecologic Cancer Intergroup Committee (GCIC) criteria; disease progression has to be radiologic or clinical; biomarker progression with CA125 after a platinum based regimen would not be sufficient evidence of disease progression; the patients must have had radiological progression to that regimen
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as > 10 mm with computed tomography (CT) scan, magnetic resonance imaging (MRI), or calipers by clinical exam
* There is no limitation in the number of prior lines of therapy
* Patients must have completed any prior chemotherapy, radiotherapy or major surgery at least 4 weeks before receiving study treatment; ongoing toxicities related to treatment must be =< grade 1 and patients with grade 2 alopecia or peripheral neuropathy can also be included; palliative radiation to < 10% of bone marrow is permissible if completed within one week of commencing study treatment as long as the toxicities secondary to palliative radiotherapy are limited to grade 1; the lesions that have received radiation treatment immediately before will be excluded as target lesions; previously irradiated lesions can be considered as targeted lesions, as long as there is prove of radiological progression
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Life expectancy of greater than 3 months
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >= 90 g/L

  * Blood transfusions are allowed at any time during the screening, treatment or follow-up period, according to the center recommendations
* Prothrombin time (PT), partial thromboplastin time (PTT) and international normalized ratio (INR) =< 1.5 upper limit of normal (ULN)
* Total bilirubin =< 1.5 x institutional upper limit of normal; unless due to Gilbert's syndrome
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 x institutional upper limit of normal (5 x if liver metastases)
* Creatinine =< 1.5 × institutional upper limit of normal OR creatinine clearance >= 40 mL/min/1.73 m^2 for patients with creatinine levels above 1.5 x institutional limit of normal
* Patients must be able to tolerate oral medication and not have evidence of active bowel obstruction

  * Note: patients can have a history of prior bowel obstruction, provided the patient is not having symptoms of bowel obstruction at the time of enrolment and the bowel obstruction is not anticipated to recur during the participation in the study
* Patients must have disease amenable to biopsy and must be willing to undergo a paired biopsy for correlative analyses (the first biopsy within 28 days prior to start of treatment and the second biopsy while on treatment)
* Women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while she is participating in this study, she should inform her treating physician immediately

  * Women of childbearing potential include women who have experienced menarche and who have not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or are not postmenopausal; postmenopause is defined as amenorrhea >= 12 consecutive months; Note: women who have been amenorrheic for 12 or more months are still considered to be of childbearing potential if the amenorrhea is possibly due to prior chemotherapy, anti-estrogens, ovarian suppression or any other reversible reason
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who previously received gemcitabine for the treatment of recurrent disease
* Patients who are receiving any other investigational agents
* Patients with clinically or radiologically unstable brain metastases are excluded from this clinical trial

  * Note: patients with stable brain metastases after treatment, for at least 3 months prior to enrolling on this trial, could participate in the study; patients should be off, or on a stable dose of steroids
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to AZD 1775 (MK-1775) or gemcitabine
* Patients taking the following prescription or non-prescription drugs or other products (i.e. grapefruit juice) are ineligible: sensitive cytochrome P450 family 3, subfamily A, polypeptide 4 (CYP3A4) substrates, CYP3A4 substrates with a narrow therapeutic index, moderate to potent inhibitors/inducers of CYP3A4; patients would be eligible if the medications can be discontinued two weeks prior to day 1 of dosing and withheld throughout the study until 2 weeks after the last dose of study medication
* Pregnant and breastfeeding women are excluded from this study
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible
* Uncontrolled intercurrent illness including, but not limited to, myocardial infarction within 6 months, congestive heart failure, symptomatic congestive heart failure, unstable angina pectoris, active cardiomyopathy, unstable ventricular arrhythmia, uncontrolled hypertension, uncontrolled psychotic disorders, serious infections, active peptic ulcer disease, active liver disease or cerebrovascular disease with previous stroke, or psychiatric illness/social situations that would limit compliance with study requirements

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2014-07-21 (Actual); Primary Completion 2022-02-03 (Actual); Study Completion 2026-02-20 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Amit M Oza, Principal Investigator — University Health Network-Princess Margaret Hospital
Locations (16):
- United States (8):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - City of Hope South Pasadena, South Pasadena, California
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
- Canada (7):
  - BCCA-Cancer Centre for the Southern Interior, Kelowna, British Columbia
  - BCCA-Vancouver Cancer Centre, Vancouver, British Columbia
  - London Regional Cancer Program, London, Ontario
  - Ottawa Hospital and Cancer Center-General Campus, Ottawa, Ontario
  - University Health Network Princess Margaret Cancer Center P2C, Toronto, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario
  - CHUM - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
- National University Hospital Singapore, Singapore, Singapore

REFERENCES:
- [Derived] Lheureux S, Cristea MC, Bruce JP, Garg S, Cabanero M, Mantia-Smaldone G, Olawaiye AB, Ellard SL, Weberpals JI, Wahner Hendrickson AE, Fleming GF, Welch S, Dhani NC, Stockley T, Rath P, Karakasis K, Jones GN, Jenkins S, Rodriguez-Canales J, Tracy M, Tan Q, Bowering V, Udagani S, Wang L, Kunos CA, Chen E, Pugh TJ, Oza AM. Adavosertib plus gemcitabine for platinum-resistant or platinum-refractory recurrent ovarian cancer: a double-blind, randomised, placebo-controlled, phase 2 trial. Lancet. 2021 Jan 23;397(10271):281-292. doi: 10.1016/S0140-6736(20)32554-X. PMID 33485453

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between Oct. 16, 2014 and Jan. 16, 2018, 124 women were enrolled, of whom 99 had high-grade serous ovarian cancer and were randomly assigned to AZD1775 plus gemcitabine (65 [66%]) or placebo plus gemcitabine (34 [34%]). 25 women with non-high-grade serous ovarian cancer were enrolled in the exploratory cohort.
Pre-assignment Details: After randomization, five patients with high-grade serous ovarian cancer were found to be ineligible (four in the experimental group and one in the control group) and did not receive treatment.
Groups:
- Arm I (WEE1 Inhibitor AZD1775, Gemcitabine Hydrochloride): Patients receive WEE1 inhibitor AZD1775 PO on days 1, 2, 8, 9, 15, and 16 and gemcitabine hydrochloride IV over 30 minutes on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
- Arm II (Placebo, Gemcitabine Hydrochloride): Patients receive placebo PO on days 1, 2, 8, 9, 15, and 16 and gemcitabine hydrochloride IV as patients in Arm I. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
- Arm III (Exploratory Cohort): Patients with non-high-grade serous ovarian cancer. Patients receive WEE1 inhibitor AZD1775 PO on days 1, 2, 8, 9, 15, and 16 and gemcitabine hydrochloride IV over 30 minutes on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Arm I (WEE1 Inhibitor AZD1775, Gemcitabine Hydrochloride) | Arm II (Placebo, Gemcitabine Hydrochloride) | Arm III (Exploratory Cohort)
Started | 65 | 34 | 25
Completed | 61 | 33 | 25
Not Completed | 4 | 1 | 0
Not completed — Adverse Event | 4 | 0 | 0
Not completed — Admission to Hospital | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm III (Exploratory WEE1 Inhibitor AZD1775, Gemcitabine: Patients with non-high-grade serous histology were enrolled in an exploratory single-arm cohort and received WEE1 inhibitor AZD1775 PO on days 1, 2, 8, 9, 15, and 16 and gemcitabine hydrochloride IV over 30 minutes on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
- Total: Total of all reporting groups
Arm/Group | Arm I (WEE1 Inhibitor AZD1775, Gemcitabine Hydrochloride) | Arm II (Placebo, Gemcitabine Hydrochloride) | Arm III (Exploratory WEE1 Inhibitor AZD1775, Gemcitabine | Total
Number analyzed (Participants) | 61 | 33 | 25 | 119
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 42 | 21 | 20 | 83
  >=65 years | 19 | 12 | 5 | 36
Age, Continuous [Median (Full Range); unit: years] | 62 [45 to 75] | 63 [43 to 76] | 58 [33 to 76] | 62 [33 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 33 | 25 | 119
  Male | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 1 | 3
  Asian | 8 | 2 | 7 | 17
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 3 | 1 | 5
  White | 48 | 27 | 16 | 91
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 0 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 38 | 25 | 12 | 75
  United States | 23 | 8 | 13 | 44

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: To evaluate the progression free survival (PFS) of subjects with recurrent platinum-resistant ovarian, fallopian tube or primary peritoneal cancer receiving gemcitabine in combination with AZD1775 compared to subjects receiving gemcitabine in combination with placebo. Progression is defined, using the Response Evaluation Criteria In Solid Tumors (RECIST v1.1) guideline, as at least a 20% increase in the sum of the diameters of target lesions or the appearance of one or more new lesions.
Time Frame: From start of treatment until date of progression or death, whichever occurs first, up to 1 year follow-up
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Arm I (WEE1 Inhibitor AZD1775, Gemcitabine Hydrochloride): Patients receive WEE1 inhibitor AZD-1775 PO on days 1, 2, 8, 9, 15, and 16 and gemcitabine hydrochloride IV over 30 minutes on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
- Arm III (Exploratory WEE1 Inhibitor AZD1775, Gemcitabine): Patients with non-high-grade serous histology were enrolled in an exploratory single-arm cohort and received WEE1 inhibitor AZD1775 PO on days 1, 2, 8, 9, 15, and 16 and gemcitabine hydrochloride IV over 30 minutes on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
Arm/Group | Arm I (WEE1 Inhibitor AZD1775, Gemcitabine Hydrochloride) | Arm II (Placebo, Gemcitabine Hydrochloride) | Arm III (Exploratory WEE1 Inhibitor AZD1775, Gemcitabine)
Number analyzed (Participants) | 61 | 33 | 25
months | 4.6 [3.6 to 6.4] | 3.0 [1.8 to 3.8] | 5.3 [1.6 to 7.7]

2. Secondary Outcome: Objective Response
Description: To evaluate the objective response per Response Evaluation Criteria in Solid Tumors (RECIST v1.1) of patients receiving gemcitabine combined with AZD1775 compared to patients receiving gemcitabine in combination with placebo. RECIST v1.1 criteria used for evaluation of target lesions: Complete Response (CR), disappearance of all target lesions; Partial Response (PR), at least a 30% decrease in the sum of the diameters of target lesions; Progressive Disease (PD), at least a 20% increase in the sum of the diameters of target lesions; Stable Disease (SD), neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD. The Best Overall Response is the best response recorded from the start of the treatment until disease progression/recurrence .
Time Frame: From start of treatment, every 6-8 weeks, until time of progression or death, whichever occurs first, up to 1 year follow-up
Measure: Count of Participants; unit: Participants
Groups:
- Arm III (Exploratory WEE1 Inhibitor AZD1775, Gemcitabine Hydrochloride): Patients with non-high-grade serous histology were enrolled in an exploratory single-arm cohort and received WEE1 inhibitor AZD1775 PO on days 1, 2, 8, 9, 15, and 16 and gemcitabine hydrochloride IV over 30 minutes on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
Arm/Group | Arm I (WEE1 Inhibitor AZD1775, Gemcitabine Hydrochloride) | Arm II (Placebo, Gemcitabine Hydrochloride) | Arm III (Exploratory WEE1 Inhibitor AZD1775, Gemcitabine Hydrochloride)
Number analyzed (Participants) | 61 | 33 | 25
Participants | 14 | 2 | 3

3. Secondary Outcome: Response According to CA125 Criteria
Description: To evaluate the GCIG CA125 response rate of patients receiving gemcitabine combined with AZD1775 compared to patients receiving gemcitabine in combination with placebo. A response according to CA-125 has occurred if there is at least a 50% reduction in CA-125 levels from a pre-treatment sample. The response must be confirmed and maintained for at least 28 days.
Time Frame: From start of treatment, every 4 weeks, until time of progression or death, whichever occurs first, up to 1 year follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (WEE1 Inhibitor AZD1775, Gemcitabine Hydrochloride) | Arm II (Placebo, Gemcitabine Hydrochloride) | Arm III (Exploratory WEE1 Inhibitor AZD1775, Gemcitabine Hydrochloride)
Number analyzed (Participants) | 61 | 33 | 25
Participants | 14 | 3 | 4

4. Secondary Outcome: Overall Survival
Description: To evaluate the overall survival of patients receiving gemcitabine combined with AZD1775 compared to patients receiving gemcitabine in combination with placebo.
Time Frame: From start of study treatment, every 12 weeks, until death, up to 22 months follow-up
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (WEE1 Inhibitor AZD1775, Gemcitabine Hydrochloride) | Arm II (Placebo, Gemcitabine Hydrochloride) | Arm III (Exploratory WEE1 Inhibitor AZD1775, Gemcitabine Hydrochloride)
Number analyzed (Participants) | 61 | 33 | 25
months | 11.4 [8.2 to 16.5] | 7.2 [5.2 to 13.2] | 13 [8.5 to 21.7]

5. Secondary Outcome: Number of Participants With Grade 3 or 4 Adverse Events Related to Study Treatment
Description: To evaluate the safety and tolerability of the combination of gemcitabine combined with AZD1775 in patients with recurrent, platinum-resistant ovarian, fallopian tube or primary peritoneal cancer.
Time Frame: From start of treatment until AE resolution, stabilization, or improvement to less than grade 2, up to 1 year follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (WEE1 Inhibitor AZD1775, Gemcitabine Hydrochloride) | Arm II (Placebo, Gemcitabine Hydrochloride) | Arm III (Exploratory WEE1 Inhibitor AZD1775, Gemcitabine Hydrochloride)
Number analyzed (Participants) | 61 | 33 | 25
Participants
  Neutropenia | 38 | 10 | 18
  Thrombocytopenia | 19 | 2 | 9
  Fatigue | 10 | 3 | 4
  Anemia | 19 | 6 | 8
  Decreased White Blood Cell Count | 33 | 6 | 16
  Decreased Lymphocyte Count | 21 | 6 | 9
  Febrile Neutropenia | 7 | 0 | 2
  Abdominal Pain | 1 | 1 | 0
  Nausea | 2 | 1 | 0
  Vomiting | 1 | 2 | 0
  Edema Trunk | 2 | 0 | 0
  Catheter Related Infection | 0 | 1 | 0
  Sepsis | 3 | 0 | 0
  Skin Infection | 0 | 1 | 0
  Urinary Tract Infection | 4 | 0 | 0
  Weight Gain | 1 | 0 | 0
  Dehydration | 1 | 1 | 2
  Hypokalemia | 6 | 0 | 2
  Hyponatremia | 0 | 1 | 0
  Hypophosphatemia | 3 | 0 | 2
  Dyspnea | 3 | 0 | 0
  Pneumonitis | 1 | 0 | 0
  Hypertension | 1 | 0 | 0
  Thromboembolic Event | 2 | 1 | 0
  Alanine Aminotransferase Increased | 2 | 2 | 0
  Aspartate Aminotransferase Increased | 3 | 3 | 0
  Diarrhea | 1 | 0 | 1
  Rash Maculo-Papular | 4 | 0 | 0
  Hypoalbuminemia | 1 | 0 | 0
  Alkaline Phosphatase Increased | 1 | 0 | 0
  Pruritis | 1 | 0 | 0
  Headache | 1 | 0 | 0
  Syncope | 1 | 0 | 0
  Anaphylaxis | 1 | 0 | 0
  Atrial Fibrillation | 1 | 0 | 0
  Pneumonia | 1 | 1 | 0
  Hematoma | 0 | 1 | 0
  Wound Complication | 0 | 1 | 0
  Fever | 0 | 0 | 1
  Enterocolitis Infection | 0 | 0 | 1
  Lung Infection | 0 | 0 | 1

6. Secondary Outcome: TP53 Mutations
Description: To evaluate TP53 mutations (presence of mutation and type of mutation) as potential predictive factors of benefit (defined as response or PFS prolongation) to AZD1775 and gemcitabine treatment. TP53 status was assessed using Sanger sequencing.
Time Frame: Baseline
Population: TP53 status was assessed in 108 patients. 8 patients had insufficient or unavailable samples and 3 patients were not tested.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (WEE1 Inhibitor AZD1775, Gemcitabine Hydrochloride) | Arm II (Placebo, Gemcitabine Hydrochloride) | Arm III (Exploratory WEE1 Inhibitor AZD1775, Gemcitabine Hydrochloride)
Number analyzed (Participants) | 56 | 33 | 19
Participants | 48 | 22 | 8

7. Secondary Outcome: p53 Protein Expression
Description: To evaluate p53 protein expression by immunohistochemistry as potential predictive factors of benefit (defined as response or PFS prolongation) to AZD1775 and gemcitabine treatment.
  Evaluating p53 expression in patients with high-grade serous ovarian cancer and in patients with high-grade serous ovarian cancer with TP53 mutations.
Time Frame: Baseline
Population: As per protocol, p53 protein expression was evaluated by immunohistochemistry to correlate with patients' mutational status of TP53
Measure: Count of Participants; unit: Participants
Groups:
- Abnormal p53 Expression in Patients With High-grade Serous Ovarian Cancer: Abnormal p53 expression in patients with high-grade serous ovarian cancer
- Abnormal p53 Expression in Patients With High-grade Serous Ovarian Cancer and With TP53 Mutations: Abnormal p53 expression in patients with high-grade serous ovarian cancer and with TP53 mutations
Arm/Group | Abnormal p53 Expression in Patients With High-grade Serous Ovarian Cancer | Abnormal p53 Expression in Patients With High-grade Serous Ovarian Cancer and With TP53 Mutations
Number analyzed (Participants) | 88 | 70
Participants | 82 | 68

8. Other Pre Specified Outcome: Patient Reported Outcomes
Description: Will be assessed using Patient Reported Outcomes-Common Terminology Criteria for Adverse Events (PRO-CTCAE).
  Each symptomatic AE is assessed with respect to 1 to 3 of the following attributes: frequency (F), severity (S) and/or interference (I) with usual or daily activities, and a recall period of 'the past 7 days'. PRO-CTCAE responses are scored from 0 to 4 with scores of 3 and 4 corresponding to high frequency, severity and/or interference. Results show the number of patients in each arm reporting high scores (3-4) for symptomatic AEs occurring in >30% of patients
Time Frame: First 3 months
Measure: Count of Participants; unit: Participants
Groups:
- Arm I (WEE1 Inhibitor AZD-1775, Gemcitabine Hydrochloride): Patients receive WEE1 inhibitor AZD-1775 PO on days 1, 2, 8, 9, 15, and 16 and gemcitabine hydrochloride IV over 30 minutes on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
- Arm III (Exploratory WEE1 Inhibitor AZD-1775, Gemcitabine): Patients with non-high-grade serous histology were enrolled in an exploratory single-arm cohort and received WEE1 inhibitor AZD-1775 PO on days 1, 2, 8, 9, 15, and 16 and gemcitabine hydrochloride IV over 30 minutes on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
Arm/Group | Arm I (WEE1 Inhibitor AZD-1775, Gemcitabine Hydrochloride) | Arm II (Placebo, Gemcitabine Hydrochloride) | Arm III (Exploratory WEE1 Inhibitor AZD-1775, Gemcitabine)
Number analyzed (Participants) | 28 | 19 | 8
Participants
  Abdominal Pain F | 10 | 9 | 1
  Abdominal Pain S | 9 | 5 | 0
  Anxiety F | 7 | 6 | 2
  Bloating F | 10 | 5 | 1
  Bloating S | 9 | 3 | 1
  Fatigue S | 16 | 6 | 4
  Fatigue I | 17 | 7 | 5

9. Other Pre Specified Outcome: TP53 Mutations in Circulating Tumor Deoxyribonucleic Acid
Description: TP53 mutations in circulating tumor deoxyribonucleic acid will be evaluated by TAm-Seq.
Time Frame: Baseline
Population: Data were not collected
Arm/Group | Arm I (WEE1 Inhibitor AZD-1775, Gemcitabine Hydrochloride) | Arm II (Placebo, Gemcitabine Hydrochloride) | Arm III (Exploratory WEE1 Inhibitor AZD-1775, Gemcitabine)
Number analyzed (Participants) | 0 | 0 | 0

10. Other Pre Specified Outcome: Change in Levels of Circulating Deoxyribonucleic Acid TP53 Mutations by TAm-Seq
Description: Levels of circulating deoxyribonucleic acid TP53 mutations will be correlated with response.
  *No results for this outcome measure
Time Frame: Baseline to up to 1 year
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Changes in pCDC2 in Skin and Tumor Tissue
Description: Validation of pCDC2 as a pharmacodynamic marker of therapy.
  *No results for this outcome measure
Time Frame: Baseline and at day 2 or 9 (course 1)
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Changes in gH2AX in Skin and Tumor Tissue
Description: Validation of gH2AX as a pharmacodynamic marker of therapy.
  *No results for this outcome measure
Time Frame: Baseline and at day 2 or 9 (course 1)
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Changes in pCDC2
Description: Changes in pCDC2 will be correlated with survival outcomes and response rate.
  *No results for this outcome measure
Time Frame: Baseline and at day 2 or 9 (course 1)
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Changes in pH2AX
Description: Changes in pH2AX will be correlated with survival outcomes and response rate.
  *No results for this outcome measure
Time Frame: Baseline and at day 2 or 9 (course 1)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse Events monitored/assessed from start of treatment until AE resolution, up to 1 year follow-up. All-Cause Mortality monitored/assessed for up to 22 months.
Description: Adverse events regularly assessed by Investigator
Arm/Group | Arm I (WEE1 Inhibitor AZD1775, Gemcitabine Hydrochloride) | Arm II (Placebo, Gemcitabine Hydrochloride) | Arm III (Exploratory WEE1 Inhibitor AZD1775, Gemcitabine Hydrochloride)
All-Cause Mortality (participants affected / at risk) | 50/61 | 30/33 | 16/25
Serious Adverse Events (participants affected / at risk) | 29/61 | 12/33 | 10/25
Other Adverse Events (participants affected / at risk) | 61/61 | 33/33 | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (WEE1 Inhibitor AZD1775, Gemcitabine Hydrochloride) (N=61) | Arm II (Placebo, Gemcitabine Hydrochloride) (N=33) | Arm III (Exploratory WEE1 Inhibitor AZD1775, Gemcitabine Hydrochloride) (N=25)
Anemia (Blood and lymphatic system disorders) | 3 (5) | 2 (3) | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 4 (5) | 0 (0) | 2 (2)
Abdominal Pain (Gastrointestinal disorders) | 4 (4) | 2 (2) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Colonic Obstruction (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Jejunal Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Obstruction Gastric (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Small Intestinal Obstruction (Gastrointestinal disorders) | 4 (5) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Edema Trunk (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1)
Fever (General disorders) | 8 (9) | 0 (0) | 0 (0)
Abdominal Infection (Infections and infestations) | 2 (3) | 0 (0) | 0 (0)
Appendicitis Perforated (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Catheter Related Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 3 (5) | 0 (0) | 0 (0)
Skin Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 4 (10) | 0 (0) | 1 (1)
Cardiac Troponin I Increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte Count Decreased (Investigations) | 1 (1) | 1 (1) | 2 (2)
Neutrophil Count Decreased (Investigations) | 7 (9) | 2 (2) | 3 (3)
Platelet Count Decreased (Investigations) | 5 (7) | 0 (0) | 1 (1)
Weight Gain (Investigations) | 1 (1) | 0 (0) | 0 (0)
White Blood Cell Decreased (Investigations) | 6 (6) | 1 (1) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Muscle Weakness Left-Sided (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary Tract Obstruction (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Right Leg Deep Vein Thrombosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Pelvic Pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 0 (0)
Treatment Hypersensitivity (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Thromboembolic Event (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Death Due to Disease Progression (General disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (WEE1 Inhibitor AZD1775, Gemcitabine Hydrochloride) (N=61) | Arm II (Placebo, Gemcitabine Hydrochloride) (N=33) | Arm III (Exploratory WEE1 Inhibitor AZD1775, Gemcitabine Hydrochloride) (N=25)
Fatigue (General disorders) | 54 (54) | 32 (32) | 20 (20)
Anemia (Blood and lymphatic system disorders) | 54 (54) | 30 (30) | 25 (25)
Nausea (Gastrointestinal disorders) | 49 (49) | 24 (24) | 20 (20)
Decreased white blood cell count (Investigations) | 54 (54) | 23 (23) | 24 (24)
Decreased platelet count (thrombocytopenia) (Investigations) | 52 (52) | 22 (22) | 21 (21)
Decreased neutrophil count (neutropenia) (Investigations) | 50 (50) | 22 (22) | 23 (23)
Decreased lymphocyte count (Investigations) | 47 (47) | 22 (22) | 20 (20)
Abdominal pain (Gastrointestinal disorders) | 45 (45) | 22 (22) | 20 (20)
Constipation (Gastrointestinal disorders) | 43 (43) | 20 (20) | 20 (20)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 42 (42) | 22 (22) | 9 (9)
Increased alanine aminotransferase (Investigations) | 39 (39) | 22 (22) | 14 (14)
Increased aspartate aminotransferase (Investigations) | 38 (38) | 23 (23) | 14 (14)
Diarrhea (Gastrointestinal disorders) | 38 (38) | 14 (14) | 12 (12)
Hypertension (Vascular disorders) | 36 (36) | 14 (14) | 8 (8)
Vomiting (Gastrointestinal disorders) | 36 (36) | 10 (10) | 12 (12)
Fever (General disorders) | 34 (34) | 14 (14) | 11 (11)
Anorexia (Metabolism and nutrition disorders) | 32 (32) | 18 (18) | 7 (7)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 30 (30) | 20 (20) | 8 (8)
Insomnia (Psychiatric disorders) | 27 (27) | 12 (12) | 10 (10)
Peripheral sensory neuropathy (Nervous system disorders) | 26 (26) | 14 (14) | 5 (5)
Hyponatremia (Metabolism and nutrition disorders) | 25 (25) | 10 (10) | 13 (13)
Back pain (Musculoskeletal and connective tissue disorders) | 24 (24) | 13 (13) | 12 (12)
Hypomagnesemia (Metabolism and nutrition disorders) | 24 (24) | 11 (11) | 6 (6)
Maculopapular rash (Skin and subcutaneous tissue disorders) | 24 (24) | 3 (3) | 11 (11)
Alopecia (Skin and subcutaneous tissue disorders) | 22 (22) | 7 (7) | 6 (6)
Chills (General disorders) | 20 (20) | 10 (10) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 20 (20) | 12 (12) | 6 (6)
Limb edema (General disorders) | 20 (20) | 12 (12) | 7 (7)
Pruritis (Skin and subcutaneous tissue disorders) | 20 (20) | 5 (5) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 19 (19) | 10 (10) | 5 (5)
Headache (Nervous system disorders) | 19 (19) | 13 (13) | 11 (11)
Hypokalemia (Metabolism and nutrition disorders) | 19 (19) | 3 (3) | 10 (10)
Weight loss (Investigations) | 19 (19) | 8 (8) | 4 (4)
Increased alkaline phosphatase (Investigations) | 18 (18) | 11 (11) | 9 (9)
Hypocalcemia (Metabolism and nutrition disorders) | 18 (18) | 7 (7) | 8 (8)
Hypophosphatemia (Metabolism and nutrition disorders) | 18 (18) | 4 (4) | 10 (10)
Anxiety (Psychiatric disorders) | 17 (17) | 9 (9) | 10 (10)
Glucose intolerance (Metabolism and nutrition disorders) | 17 (17) | 10 (10) | 5 (5)
Abdominal distension (Gastrointestinal disorders) | 12 (12) | 13 (13) | 4 (4)
Bloating (Gastrointestinal disorders) | 12 (12) | 11 (11) | 7 (7)
Thromboembolic event (Vascular disorders) | 10 (10) | 7 (7) | 5 (5)
Febrile neutropenia (Blood and lymphatic system disorders) | 10 (10) | 7 (7) | 5 (5)
Dehydration (Metabolism and nutrition disorders) | 6 (6) | 2 (2) | 6 (6)
Dizziness (Nervous system disorders) | 15 (15) | 5 (5) | 6 (6)
Oral mucositis (Gastrointestinal disorders) | 15 (15) | 3 (3) | 3 (3)
Urinary tract infection (Infections and infestations) | 14 (14) | 3 (3) | 3 (3)
Urinary frequency (Renal and urinary disorders) | 12 (12) | 3 (3) | 3 (3)
Dysgeusia (Nervous system disorders) | 12 (12) | 6 (6) | 1 (1)
Ascites (Gastrointestinal disorders) | 12 (12) | 9 (9) | 4 (4)
Dry mouth (Gastrointestinal disorders) | 9 (9) | 0 (0) | 0 (0)
Pain (General disorders) | 9 (9) | 0 (0) | 0 (0)
Increased creatinine (Investigations) | 9 (9) | 6 (6) | 2 (2)
Depression (Psychiatric disorders) | 9 (9) | 6 (6) | 7 (7)
Myalgia (Musculoskeletal and connective tissue disorders) | 8 (8) | 6 (6) | 5 (5)
Acneiform rash (Skin and subcutaneous tissue disorders) | 8 (8) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 8 (8) | 3 (3) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 2 (2) | 6 (6)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 8 (8) | 4 (4) | 5 (5)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 8 (8) | 3 (3) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 7 (7) | 3 (3) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 7 (7) | 7 (7) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 7 (7) | 0 (0) | 3 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 3 (3) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 4 (4) | 3 (3)
Weight gain (Investigations) | 7 (7) | 4 (4) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (6) | 5 (5) | 1 (1)
Flatulence (Gastrointestinal disorders) | 6 (6) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 6 (6) | 3 (3) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (6) | 5 (5) | 1 (1)
Urinary urgency (Renal and urinary disorders) | 6 (6) | 3 (3) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 6 (6) | 4 (4) | 2 (2)
Flu like symptoms (General disorders) | 6 (6) | 5 (5) | 4 (4)
Urinary tract obstruction (Renal and urinary disorders) | 6 (6) | 1 (1) | 3 (3)
Blurred vision (Eye disorders) | 5 (5) | 4 (4) | 4 (4)
Peripheral motor neuropathy (Nervous system disorders) | 5 (5) | 3 (3) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 5 (5) | 3 (3) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 5 (5) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 4 (4) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 5 (5) | 2 (2) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 5 (5) | 3 (3) | 2 (2)
Bruising (Injury, poisoning and procedural complications) | 4 (4) | 1 (1) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 4 (4) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 4 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (4) | 4 (4) | 4 (4)
Non-cardiac chest pain (General disorders) | 4 (4) | 4 (4) | 2 (2)
Vaginal hemorrhage (Reproductive system and breast disorders) | 4 (4) | 1 (1) | 4 (4)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 0 (0)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Hot flashes (Vascular disorders) | 3 (3) | 5 (5) | 2 (2)
Memory impairment (Nervous system disorders) | 3 (3) | 2 (2) | 2 (2)
Pelvic pain (Reproductive system and breast disorders) | 3 (3) | 5 (5) | 3 (3)
Tinnitus (Ear and labyrinth disorders) | 3 (3) | 2 (2) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 3 (3) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1) | 0 (0)
Increase blood bilirubin (Investigations) | 3 (3) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 3 (3) | 0 (0) | 1 (1)
Malaise (General disorders) | 3 (3) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 3 (3) | 0 (0) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 3 (3) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 3 (3) | 3 (3) | 5 (5)
Phlebitis (Vascular disorders) | 3 (3) | 2 (2) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 2 (2)
Skin infection (Infections and infestations) | 2 (2) | 6 (6) | 3 (3)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2) | 3 (3) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 3 (3)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 2 (2)
Nail discoloration (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Localized edema (General disorders) | 2 (2) | 2 (2) | 3 (3)
Lymphedema (Vascular disorders) | 0 (0) | 2 (2) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1)
Hematoma (Vascular disorders) | 1 (1) | 2 (2) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 3 (3)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 3 (3)
Increased lymphocyte count (Investigations) | 1 (1) | 0 (0) | 3 (3)
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 (1) | 0 (0) | 2 (2)
Injection site reaction (General disorders) | 1 (1) | 0 (0) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2)
Vaginal infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Mucosal infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
* Randomization in a 2:1 ratio is associated with reduced statistical power - increased the sample size by 12% compared to a 1:1 randomization design
* No stratification factors because of the small sample size, potentially resulting in imbalances in BRCA mutation status
* Absence of quality-of-life assessment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-03): https://cdn.clinicaltrials.gov/large-docs/75/NCT02101775/Prot_SAP_000.pdf